CLINICAL TRIAL: NCT03687879
Title: Women's Evaluation of the Childbirth Experience: From Pregnancy to Postpartum
Acronym: EVA (ECE)
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0172
Record Dates: First submitted 2018-09-21; First posted 2018-09-27 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Childbirth Problems; Pregnancy Related; Behavior Problem
MeSH Terms: conditions — Mental Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — Reporting of medical gestures or acts, speech, embarrassing or hurtful attitudes during pregnancy follow-up or during hospitalization outside childbirth, or during childbirth or immediate after birth among women giving birth in one of the 26 maternity hospitals in the period of observation period.

SUMMARY:
Women report inappropriate health professional behaviour towards them during pregnancy or childbirth on social networks. However, to date, no data are available to estimate the number of women concerned. These data are necessary to characterize these behaviours to get out of this polemic and build a reflection on the improvement of the patient relationship and the emotional security of women.

ELIGIBILITY:
Inclusion Criteria:

* major women
* who understand french language

Exclusion Criteria:

* Women refusing to participate
* having given birth at home
* whose fetus or newborn has died

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All women having given birth of a living child, whatever the term, on 1 week of observation in one of the 26 maternity units participating .
Sampling Method: Non-Probability Sample
Enrollment: 799 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2019-01-13 (Actual)

PRIMARY OUTCOMES:
Proportion of women reporting inappropriate behavior | about 1 week
  An inappropriate behavior, also called "obstetric violence" is defined by medical gestures or acts, speech, embarrassing or hurtful attitudes during pregnancy follow-up or during hospitalization outside childbirth, or during childbirth or immediate after birth.
  Womens will compleat a questionnaire to report this inappropriate behavior at the exit of the maternity.
Proportion of women reporting inappropriate behavior | at 2 months
  An inappropriate behavior, also called "obstetric violence" is defined by medical gestures or acts, speech, embarrassing or hurtful attitudes reported by womens with a questionnaire 2 months after exit of the maternity.

CONTACTS AND LOCATIONS:
Locations (26):
- France (26):
  - Hôpital Privé d'Ambérieu, Ambérieu-en-Bugey
  - Polyclinique du Beaujolais, Arnas
  - CH d'ARDECHE MERIDIONALE, Aubenas
  - CH de BOURG EN BRESSE - Pôle Mère Enfant, Bourg-en-Bresse
  - Centre Hospitalier Pierre Oudot, Bourgoin
  - Clinique St Vincent de Paul, Bourgoin
  - Hôpital Femme Mère Enfant, Bron
  - Clinique du Val D'ouest, Écully
  - Centre Hospitalier de Givors, Givors
  - Centre Hospitalier de Villefranche Sur Saône Hôpital Nord-Ouest, Gleizé
  - Hôpital Privé Drôme Ardèche Clinique Pasteur, Guilherand-Granges
  - Réseau AURORE, service de gynécologie Obstétrique, Hôpital de la Croix-Rousse, Lyon
  - Centre Hospitalier St Joseph St Luc, Lyon
  - Hôpital Prive Natecia, Lyon
  - Hôpital de La Croix-Rousse, Lyon
  - Ch Montelimar Ghpp, Montélimar
  - CH du HAUT-BUGEY, Oyonnax
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Polyclinique Lyon Nord Service Maternité (NATECIA), Rillieux-la-Pape
  - Hôpitaux Drôme Nord - Site de Romans, Romans-sur-Isère
  - Centre Hospitalier de Sainte Foy les Lyon, Sainte-Foy-lès-Lyon
  - Centre Hospitalier de Valence, Valence
  - Clinique de l'Union, Vaulx-en-Velin
  - Ghm Les Portes Du Sud, Vénissieux
  - Ch Vienne Lucien Hussel, Vienne
  - Clinique du Tonkin, Villeurbanne

IPD SHARING:
Plan to Share IPD: No